CLINICAL TRIAL: NCT00795379
Title: Testing the Use of Interoceptive Exposure to Reduce Barriers to Psychotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: G.V. (Sonny) Montgomery VA Medical Center (U.S. Federal Agency)
Responsible Party: Kevin S. Del Ben, Ph.D. Assistant Professor, G.V. (Sonny) Montgomery VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRECC 5-1006
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Anxiety
Keywords: Psychotherapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IE (Experimental): Participants will complete an at home four-week, intervention targeting their negative cognitions triggered by physical sensations. The goal of IE is to purposefully induce bodily sensations related to autonomic arousal so that participants can learn that those sensations are not harmful. IE and Cognitive restructuring have been found to be superior to progressive muscle relaxation as a way to avoid aversive autonomic sensations.
  Interventions: Behavioral: Interoceptive Exposure
- 2 (No Intervention): waitlist control

INTERVENTIONS:
Behavioral: Interoceptive Exposure — Exposure to internal stimuli.
  Arms: IE

SUMMARY:
To assess the effectiveness of Interoceptive Exposure (IE) as a treatment to reduce negative cognitions and arousal in a veteran sample during an anxiety-inducing situation (i.e., the Trier Social Stressor Task - an analogue to the anxiety of undergoing exposure-based treatment). After completing the initial screening, qualifying participants will complete a pre-intervention assessment at UMC (structured clinical interview, self-report measures, and a treatment-engagement analogue exercise). Half of the participants will be randomized into either supportive counseling or to the treatment protocol at GVSMVAMC consisting of four sessions of Interoceptive Exposure over a four week period targeting interoceptive stimuli. Veterans will be assessed a second time at UMC after treatment (5 to 6 weeks after the first assessment). Participants will include approximately 40 male OEF/OIF veterans with combat-related PTSD recruited from the Trauma Recovery Program (TRP) and Post-deployment Clinic at the G.V. (Sonny) Montgomery VAMC (GVSMVAMC). Following the pre-intervention assessment, veterans will be randomized into one of two groups. Half of the veterans (n = 20) will receive received four weeks of supportive counseling while the other half will receive four weeks of Interoceptive Exposure (IE). The proposed study examines anxiety sensitivity (AS) as a possible barrier to treatment engagement in exposure therapy for PTSD. AS is a dispositional cognitive characteristic defined as the fear of sensations directly related to autonomic arousal that arises from the belief that these sensations have harmful consequences. Interoceptive Exposure (IE) is an intervention that: 1) helps individuals with high AS increase their tolerance to the somatic sensations of arousal; and 2) promotes an adaptive appraisal of fear-related sensations The current study will use a social stressor task to assess the affect of IE on AS and avoidance among veterans who have PTSD, thereby increasing the likelihood that a veteran will enter into, and remain in, treatment for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Interested OEF/OIF veterans with a reported history of combat-related trauma, probable PTSD diagnosis (score above 44 on the PTSD Checklist), scores above 28 on the Anxiety Sensitivity Index (ASI), and who have been medically cleared will be invited to participate (study personnel will assist the participant in getting clearance from their primary care physician or TRP staff).

Exclusion Criteria:

* Veterans will be excluded if they are judged to have medical conditions that might limit cooperation or compromise the integrity of the self-report or psychophysiological data (e.g., uncontrolled blood pressure, severe asthma, dementia, psychotic disorder, acute mania, current substance abuse, or taking medications that would reduce physiological responding). Veterans who are currently receiving (or who are scheduled to begin) individual exposure-based treatment for PTSD will be excluded from the study. As this project is designed as a pilot study, no exclusions will be made based on previous treatment or previous treatment refusal; however, treatment history data will be collected.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- G.V. (Sonny) Montgomery VAMC, Jackson, Mississippi, United States